CLINICAL TRIAL: NCT03966417
Title: Exercise Training After Transcatheter Aortic Valve Implantation
Acronym: FitTAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, prof. Borut Jug, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLFitTAVI
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Aortic Valve Stenosis; TAVI; Transcatheter Aortic Valve Implantation; Rehabilitation
Keywords: exercise training
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Active Comparator): Patient to be randomized to "exercise training group" will have exercise training sessions 2 times per week for a period of 12 weeks. They will undergo moderate continuous exercise training at 75% of Vo2max.
  Interventions: Other: Exercise training
- Usual care group (No Intervention): Patient to be randomized to "usual care group" will undergo standard care fo 12 weeks.

INTERVENTIONS:
Other: Exercise training — Continuous exercise training 2 times per week for a period of 12 weeks.
  Other Names: Rehabilitation
  Arms: Exercise training group

SUMMARY:
In this prospective, controlled trial, patient after TAVI will be randomized to either exercise training or usual care group.

DETAILED DESCRIPTION:
Patients after transcatheter aortic valve replacement (TAVI) are particularly old and severely deconditioned and are thus likely to benefit from cardiac rehabilitation programs. In this controlled trial, patients after TAVI will be randomized to either exercise training or usual care.

The aim of our study is to compare the effect of exercise training vs. usual care on:

1. exercise capacity
2. vascular function
3. parameters of heart failure, inflammation and homeostasis
4. arrhythmogenic potential
5. health-related quality of life

ELIGIBILITY:
Inclusion Criteria:

* TAVI procedure 3-6 months prior to inclusion,
* movability (100 meters or more on 6-minute walking test after TAVI),
* ability to attend a 12 week exercise training program,
* physical and clinical ability to attend the rehabilitation program at the discretion of the researcher,
* optimal medical treatment,
* pre-signed statement of a conscious and free consent to the inclusion in the clinical trial.

Exclusion Criteria:

* contraindications for exercise training,
* unstable hearth (uncontrollable heart failure - New York Heart Association stage IV, dysrhythmias, uncontrollable myocardial ischemia),
* patient's decision to undergo TAVI despite receiving a recommendation for Surgical Aortic Valve Repair by the heart team,
* non-cardiac physical impairment that would prevent exercise training on stationary bike,
* uncontrolled pulmonary disease (FEV1 <50%),
* echocardiographic signs of prosthesis dysfunction according to the Valve Academic Research Consortium (valve orifice area of b1.2 cm2 plus a mean transaortic pressure gradient of ≥20 mm Hg, or a velocity of ≥3 m/s, at least moderate paravalvular regurgitation),
* TAVI access site complication,
* important peripheral vascular disease, musculoskeletal disease or central nervous system disease, which prevents exercise training on stationary bike,
* recent (less than 3 months) acute events or illnesses that are contraindications for exercise training.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change of maximal oxygen uptake during exercise | 3 months
  ml/kg/min

SECONDARY OUTCOMES:
Change of flow-mediated dilatation (FMD) of the brachial artery | 3 months
  % flow-mediated dilatation and arterial stiffness
Change of arterial stiffness coefficient | 3 months
  coefficient
Change of value of blood N terminal-proBNP | 3 months
  ng/l
Change of value of blood D-dimer | 3 months
  microg/l
Change of value from-the-questionnaire-obtained quality of life | 3 months
  points
Change of ECG waves | 3 months
  Estimated with digital high-resolution ECG
Change in the result of the 6-minute walking test | 3 months
  metres
Change og the heart rate variability | 3 months
  Estimated with digital high-resolution ECG

OTHER OUTCOMES:
Change of heart rate recovery | 3 months
  beats/min

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, MD, PhD, Principal Investigator — University Medical Centre Ljubljana, Slovenia
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chakos A, Wilson-Smith A, Arora S, Nguyen TC, Dhoble A, Tarantini G, Thielmann M, Vavalle JP, Wendt D, Yan TD, Tian DH. Long term outcomes of transcatheter aortic valve implantation (TAVI): a systematic review of 5-year survival and beyond. Ann Cardiothorac Surg. 2017 Sep;6(5):432-443. doi: 10.21037/acs.2017.09.10. PMID 29062738
- [Background] Pressler A, Christle JW, Lechner B, Grabs V, Haller B, Hettich I, Jochheim D, Mehilli J, Lange R, Bleiziffer S, Halle M. Exercise training improves exercise capacity and quality of life after transcatheter aortic valve implantation: A randomized pilot trial. Am Heart J. 2016 Dec;182:44-53. doi: 10.1016/j.ahj.2016.08.007. Epub 2016 Aug 26. PMID 27914499
- [Background] Dalal HM, Doherty P, Taylor RS. Cardiac rehabilitation. BMJ. 2015 Sep 29;351:h5000. doi: 10.1136/bmj.h5000. No abstract available. PMID 26419744
- [Background] McMahon SR, Ades PA, Thompson PD. The role of cardiac rehabilitation in patients with heart disease. Trends Cardiovasc Med. 2017 Aug;27(6):420-425. doi: 10.1016/j.tcm.2017.02.005. Epub 2017 Feb 15. PMID 28318815
- [Background] Butchart EG, Gohlke-Barwolf C, Antunes MJ, Tornos P, De Caterina R, Cormier B, Prendergast B, Iung B, Bjornstad H, Leport C, Hall RJ, Vahanian A; Working Groups on Valvular Heart Disease, Thrombosis, and Cardiac Rehabilitation and Exercise Physiology, European Society of Cardiology. Recommendations for the management of patients after heart valve surgery. Eur Heart J. 2005 Nov;26(22):2463-71. doi: 10.1093/eurheartj/ehi426. Epub 2005 Aug 15. PMID 16103039
- [Background] Voller H, Salzwedel A, Nitardy A, Buhlert H, Treszl A, Wegscheider K. Effect of cardiac rehabilitation on functional and emotional status in patients after transcatheter aortic-valve implantation. Eur J Prev Cardiol. 2015 May;22(5):568-74. doi: 10.1177/2047487314526072. Epub 2014 Feb 27. PMID 24577878
- [Background] Russo N, Compostella L, Tarantini G, Setzu T, Napodano M, Bottio T, D'Onofrio A, Isabella G, Gerosa G, Iliceto S, Bellotto F. Cardiac rehabilitation after transcatheter versus surgical prosthetic valve implantation for aortic stenosis in the elderly. Eur J Prev Cardiol. 2014 Nov;21(11):1341-8. doi: 10.1177/2047487313494029. Epub 2013 Jun 11. PMID 23757283
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483